CLINICAL TRIAL: NCT03612375
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Oxidative Stress Substudy of ESTxENDS
Brief Title: ESTxENDS Trial-Substudy on Oxidative Stress Induced by Electronic Nicotine Delivery Systems (ENDS) Measured in Urine
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332c
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Oxidative Stress
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Oxidative stress outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking.

Smoking induces inflammation leading to acute and chronic oxidative stress, both evidenced in in vitro and in vivo studies. Tobacco-smoke contains free reactive radicals that generate reactive oxygen species (ROS). Afterwards ROS in turn induce oxidative stress, which likely plays a key role in causing airways and related pathologies linked to tobacco-smoke exposure. Acute and chronic oxidative stress can be measured by quantifying two biomarkers in urine samples: 8-iso-prostaglandin F2α (8-isoprostane) and 8-Oxo-2'-deoxyguanosine (8-OHdG). 8-isoprostane, a marker of lipoperoxidation, results mainly from the non-enzymatic action of free radical attack on arachidonic fatty acids. 8-OHdG is a marker of DNA oxidation caused by ROS, and a predictor of lung cancer.

Oxidative stress between smokers who quit (with or without ENDS) and those who use ENDS for a long time have not yet been assessed in the setting of a randomized controlled trial (RCT). This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events, the exposure to inhaled chemicals and the effect of ENDS on health-related outcomes, in particular by measuring oxidative stress in urine samples.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Measures of oxidative stress by means of exhaled breath condensates and urine samples will be assessed at baseline and at 6-, 12- and 24- months' follow-up.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Persons having used ENDS regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other drug therapy helping smokers quit (varenicline, bupropion) within the 3 months preceding the baseline visit
* Plans to move out of the country within the next 6 months, or cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Urinary 8-OHdG concentrations to asses oxidative stress_1 | 6 months post quit date
  Oxidative stress assessed by 8-OHdG concentrations in urine.
Urinary 8-OHdG concentrations to asses oxidative stress_2 | 12 months post quit date
  Oxidative stress assessed by 8-OHdG concentrations in urine.
Urinary 8-OHdG concentrations to asses oxidative stress_3 | 24 months post quit date
  Oxidative stress assessed by 8-OHdG concentrations in urine.
Urinary 8-isoprostane concentrations to asses oxidative stress_1 | 6 months post quit date
  Oxidative stress assessed by 8-isoprostane concentrations in urine.
Urinary 8-isoprostane concentrations to asses oxidative stress_2 | 12 months post quit date
  Oxidative stress assessed by 8-isoprostane concentrations in urine.
Urinary 8-isoprostane concentrations to asses oxidative stress_3 | 24 months post quit date
  Oxidative stress assessed by 8-isoprostane concentrations in urine.

SECONDARY OUTCOMES:
Change in urinary 8-OHdG concentrations to asses oxidative stress | Change from baseline to 6,12, 24 months post quit date
  Oxidative stress assessed by 8-OHdG concentrations in urine.
Change in urinary 8-isoprostane concentrations to asses oxidative stress | Change from baseline to 6,12, 24 months post quit date
  Oxidative stress assessed by 8-isoprostane concentrations in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] van der Vaart H, Postma DS, Timens W, ten Hacken NH. Acute effects of cigarette smoke on inflammation and oxidative stress: a review. Thorax. 2004 Aug;59(8):713-21. doi: 10.1136/thx.2003.012468. PMID 15282395
- [Background] Pryor WA, Stone K. Oxidants in cigarette smoke. Radicals, hydrogen peroxide, peroxynitrate, and peroxynitrite. Ann N Y Acad Sci. 1993 May 28;686:12-27; discussion 27-8. doi: 10.1111/j.1749-6632.1993.tb39148.x. No abstract available. PMID 8512242
- [Background] Yamaguchi Y, Nasu F, Harada A, Kunitomo M. Oxidants in the gas phase of cigarette smoke pass through the lung alveolar wall and raise systemic oxidative stress. J Pharmacol Sci. 2007 Mar;103(3):275-82. doi: 10.1254/jphs.fp0061055. Epub 2007 Mar 2. PMID 17332694
- [Background] Hartmann-Boyce J, McRobbie H, Bullen C, Begh R, Stead LF, Hajek P. Electronic cigarettes for smoking cessation. Cochrane Database Syst Rev. 2016 Sep 14;9(9):CD010216. doi: 10.1002/14651858.CD010216.pub3. PMID 27622384
- [Background] Campos C, Guzman R, Lopez-Fernandez E, Casado A. Urinary biomarkers of oxidative/nitrosative stress in healthy smokers. Inhal Toxicol. 2011 Feb;23(3):148-56. doi: 10.3109/08958378.2011.554460. PMID 21391783
- [Background] Haswell LE, Papadopoulou E, Newland N, Shepperd CJ, Lowe FJ. A cross-sectional analysis of candidate biomarkers of biological effect in smokers, never-smokers and ex-smokers. Biomarkers. 2014 Aug;19(5):356-67. doi: 10.3109/1354750X.2014.912354. Epub 2014 May 22. PMID 24854418
- [Background] Lowe FJ, Gregg EO, McEwan M. Evaluation of biomarkers of exposure and potential harm in smokers, former smokers and never-smokers. Clin Chem Lab Med. 2009;47(3):311-20. doi: 10.1515/CCLM.2009.069. PMID 19676143
- [Background] Basu S. F2-isoprostanes in human health and diseases: from molecular mechanisms to clinical implications. Antioxid Redox Signal. 2008 Aug;10(8):1405-34. doi: 10.1089/ars.2007.1956. PMID 18522490
- [Background] Morrow JD, Roberts LJ 2nd. The isoprostanes. Current knowledge and directions for future research. Biochem Pharmacol. 1996 Jan 12;51(1):1-9. doi: 10.1016/0006-2952(95)02072-1. PMID 8534261
- [Background] Seet RC, Lee CY, Loke WM, Huang SH, Huang H, Looi WF, Chew ES, Quek AM, Lim EC, Halliwell B. Biomarkers of oxidative damage in cigarette smokers: which biomarkers might reflect acute versus chronic oxidative stress? Free Radic Biol Med. 2011 Jun 15;50(12):1787-93. doi: 10.1016/j.freeradbiomed.2011.03.019. Epub 2011 Mar 17. PMID 21420490
- [Background] Wu LL, Chiou CC, Chang PY, Wu JT. Urinary 8-OHdG: a marker of oxidative stress to DNA and a risk factor for cancer, atherosclerosis and diabetics. Clin Chim Acta. 2004 Jan;339(1-2):1-9. doi: 10.1016/j.cccn.2003.09.010. PMID 14687888
- [Background] Lowe FJ, Luettich K, Gregg EO. Lung cancer biomarkers for the assessment of modified risk tobacco products: an oxidative stress perspective. Biomarkers. 2013 May;18(3):183-95. doi: 10.3109/1354750X.2013.777116. Epub 2013 Mar 27. PMID 23530763